CLINICAL TRIAL: NCT04376801
Title: A Retrospective Study on the Outcome of Different Fixation Methods After Olecranon Osteotomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Chen chen, Resident, Beijing Jishuitan Hospital
Other Study IDs: 201708-05
Record Dates: First submitted 2020-01-25; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Distal Humerus Fractures; Osteotomy; Fixation Device; Complications
Keywords: Distal Humerus Fractures; Olecranon Osteotomy; Plate Fixation; Tension-band Fixation
MeSH Terms: conditions — Humeral Fractures, Distal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tension-band Fixation Group: Patients with distal humerus fractures admitted to our hospital in 2012-2017 who had been performed open reduction and internal fixation through olecranon osteotomy approach were selected. All patients were devided into two groups by different fixation method. Patients who had been performed tension-band fixation after olecranon osteotomy were classified into Tension-band Fixation Group.
- Plate Fixation Group: Patients with distal humerus fractures admitted to our hospital in 2012-2017 who had been performed open reduction and internal fixation through olecranon osteotomy approach were selected. All patients were devided into two groups by different fixation method. Patients who had been performed plate fixation after olecranon osteotomy were classified into Plate Fixation Group.

SUMMARY:
Humeral intercondylar fractures are very challenging in clinical treatment. There are many problems not clear. One of the important problems remained to be solved is which fixation method can achieve the best effects after olecranon osteotomy. Therefore, the investigators are going to perform a retrospective analysis of patients with distal humerus fractures admitted to their hospital in 2012-2017 to compare the functional outcomes of elbow joints with tension-band fixation and plate fixation after olecranon osteotomy.

DETAILED DESCRIPTION:
Humeral intercondylar fractures are very challenging in clinical treatment. Because the humeral intercondylar fracture is comminuted and often occurs in elderly patients with osteoporosis, it is difficult to achieve rigid fixation during the operation and failure of fixation occurs from time to time after the operation. Nonunion and reoperation have brought great sufferings to the patients.In recent years, both surgical methods and technique of internal fixation have been greatly improved, but there are still many problems not clear. Olecranon osteotomy has been proven to be an effective approach for comminuted intercondylar fractures and there are different fixation methods to fix the proximal ulna after intercondylar fixation. However, it is not clear which method can achieve the best effects. Therefore, the investigators are going to perform a retrospective analysis of patients with distal humerus fractures admitted to their hospital in 2012-2017 to compare the functional outcomes of elbow joints with tension-band fixation and plate fixation after olecranon osteotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old;
2. Distal humerus fractures.

Exclusion Criteria:

1. Pathological fractures;
2. Combined with fractures of ipsilateral upper limb;
3. Fracture over 2 weeks;
4. Patients who refused surgical treatment;
5. Patients who were unable to obtain the 1 year follow-up data after the operation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were operated in our hospital because of distal humerus fractures in 2012-2017.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional result of elbow (objective) | 1 year post-op
  Assess function of patients' affected elbow by MEPS (Mayo elbow performance score)
Functional result of elbow (subjective) | 1 year post-op
  Assess function of patients' affected elbow by and DASH (Disabilities of arm, shoulder and hand)
Range of motion of elbow | 1 year post-op
  Measure and record the ROM of the affected elbow，including flexion, extension, pronation and supination degree.

SECONDARY OUTCOMES:
Complication: infection | 1 year post-op
  Record patients' information about infection if any, including superficial and deep infection.
Complication:stiffness | 1 year post-op
  Record whether the patients had elbow stiffness (ROM<100° or arthrolysis having been performed)
Complication: internal fixation irritation | 1 year post-op
  Record whether there were internal fixation irritations
Complication: failure of internal fixation | 1 year post-op
  Record whether the patients have gone through internal fixation failure
Complication: post-traumatic arthritis | 1 year post-op
  Record if the patients have developed into post-traumatic arthritis, if any, record the degree.
severity of ulnar nerve injury | 1 year post-op
  Assess and record severity of ulnar nerve injury (paralysis or weakness of intrinsic muscle of hand or parathesia of ring and little finger)
severity of pain | 1 year post-op
  Assess severity of pain by VAS (Visual analogue scale)
nounion | 1 year post-op
  Record if there is nonunion of the olecranon (evaluated by X-ray or CT scan)

CONTACTS AND LOCATIONS:
Overall Officials: Xieyuan Jiang, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, China